CLINICAL TRIAL: NCT06556927
Title: Effect of Laughter Yoga on Stress and Quality of Life in Pregnant Women With Gestational Diabetes
Brief Title: The Laughter, Pregnancy, Anxiety and Llife Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Ayca Solt Kirca, Asssociate professor, Kırklareli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KırklareliAS-12
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Life Style; Gestational Diabetes; Pregnancy Related
Keywords: Pregnancy; Gestational Diabetes; Laughter yoga
MeSH Terms: conditions — Anxiety Disorders; Diabetes, Gestational | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter yoga group (Experimental): Laughter yoga will be performed in 8 sessions, 2 days a week for 4 weeks. The duration of each session will be 40 minutes. Laughter yoga sessions will be held on a day suitable for all participants and with the participation of at least 8 people. The session will start with warm-up exercises and continue with laughter exercises. People in the group will do these exercises with the guidance of the researcher.
  Interventions: Other: Laughter yoga
- Control group (No Intervention): Participants in this group will consist of people who do not routinely do any practice on their own to reduce anxiety and increase life quality. The researcher will ask the participants via phone 4 times a week for 1 month whether they have taken any action to reduce their anxiety and increase life quality symptoms.
  Participants who use any of the pharmacological or non-pharmacological practices to reduce anxiety and increase life quality symptoms will be excluded from the study.

INTERVENTIONS:
Other: Laughter yoga — Part 1: Deep Breathing Exercises: Raise the arms up towards the sky and take a deep breath as possible and hold the breath for 4-5 seconds. This application is repeated several times. This section takes approximately 5-10 minutes.
  Part 2: Warm-up exercises: Hands are kept parallel to each other and clapped. The tips of the fingers and palms touch each other, the acupuncture points on both hands are stimulated and the individual's energy level increases.
  Section 3: Childish Games: In this section there are childish games. These games are visualized in the mind and the participants are asked to raise their arms upwards in the shape of the letter "Y".This section takes approximately 10 minutes.
  Section 4: Laughter Exercises: Participants are given verbal guidance such as "Put your hand on your heart, feel your heartbeat, let's exhale with a smile, let's make a wish or pray" and the laughter exercise is terminated. This section takes approximately 15 minutes.
  Arms: Laughter yoga group

SUMMARY:
Gestational Diabetes is one of the most common medical complications during pregnancy. It is seen between the 24th and 28th weeks of pregnancy with the increase in insulin resistance in the second trimester and ends with the end of the birth process. Due to this feature, it is distinguished from Type 2 diabetes. This disease, which is seen for the necessary energy needs of the fetus and placenta, is defined as the diabetogenic effect of pregnancy.

Laughter is a universal response to humorous stimuli that exists in our lives. Laughter yoga is holistic with breathing techniques. It is a form of yoga that utilizes the brain's inability to distinguish between real and fake laughter. Laughter yoga helps people cope with stressful times and helps the person control themselves by reducing negative cognitive reactions. In line with this information, the aim of the study was to determine the effect of laughter yoga applied to pregnant women with gestational diabetes on perceived stress and quality of life.

DETAILED DESCRIPTION:
Gestational Diabetes is one of the most common medical complications during pregnancy. It is seen between the 24th and 28th weeks of pregnancy with the increase in insulin resistance in the second trimester and ends with the end of the birth process. Due to this feature, it is distinguished from Type 2 diabetes. This disease, which is seen for the necessary energy needs of the fetus and placenta, is defined as the diabetogenic effect of pregnancy.

The American College of Obstetricians and Gynecologists (ACOG) defines GDM as "abnormal glucose tolerance that begins in pregnancy or is first diagnosed during pregnancy." However, the American Diabetes Association (ADA) and the World Health Organization (WHO) want to distinguish cases with possible diabetes diagnosed before pregnancy and diagnosed during pregnancy from glucose intolerance that occurs as a result of pregnancy and is related to pregnancy. Laughter is a universal response to humorous stimuli that exists in our lives. Laughter yoga is holistic with breathing techniques. It is a form of yoga that utilizes the brain's inability to distinguish between real and fake laughter. Laughter yoga helps people cope with stressful times and helps the person control themselves by reducing negative cognitive reactions. Laughter yoga is a non-pharmacological and non-invasive alternative treatment method. Laughter yoga is a type of communication that combines pleasant emotions, smiles, and laughter. It is a different approach from medical treatments; indicates that the psychological aspects of the brain must change in order for both the mind and body to be healthy. Maternal complications increase in pregnant women diagnosed with gestational diabetes. The prospective psychological concerns experienced by the pregnant woman (low risk, preterm birth, low birth weight) negatively affect the quality of life of the pregnant woman. In line with this information, the aim of the study was to determine the effect of laughter yoga applied to pregnant women with gestational diabetes on perceived stress and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Answering the survey and scale forms completely
* Being 18 years of age or older
* Being able to read and understand Turkish
* Not having any physical or mental problems that would prevent communication
* Pregnant women diagnosed with gestational diabetes
* Being in social media accounts and WhatsApp groups
* Scoring 35 and above on the STAI scale
* Scoring 37 and above on the quality of life scale during pregnancy

Exclusion Criteria:

* Not volunteering to participate in the study
* Incomplete responses to surveys and scales
* Being under the age of 18
* Not understanding Turkish
* Having any physical or mental problems that would prevent communication
* Pregnant women who have not been diagnosed with gestational diabetes

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 80 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale During Pregnancy | between 2 to 4 weeks
  It aims to optimally evaluate the quality of life of women with normal pregnancies and consists of nine items. It is a scale specific to singleton pregnancies that should be used in clinical and social research because it provides a better perspective on the quality of life of pregnant women rather than a general quality of life scale. The total score of the scale varies between 9-45, with higher scores indicating higher quality of life.There is no adverse substance in the scale. It can be used in every trimester
State-Trait Anxiety Inventory | between 2 to 4 weeks
  The lowest and highest scores that can be obtained from each subscale are 20 and 80, respectively. Higher scores are associated with more anxiety.
Psychometric Properties of Eurohis (Whoqol-8.Tr) Turkish Version in Turkish Society | between 2 to 4 weeks
  EUROHIS-QOL 8 was developed by the World Health Organization (WHO) in 2003. It consists of 8 items and was validated in Turkish by Eser et al in 2010. The total score determines the overall quality of life level; higher scores indicate higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: AYCA SOLT KIRCA, Phd, Study Chair — Kırklareli University
Locations (1):
- Kırklareli University, Kırklareli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No